CLINICAL TRIAL: NCT03053089
Title: A Two-Stage, Phase 1/2, Open-Label Study of the Human Insulin Receptor Monoclonal Antibody-Human Alpha-L-iduronidase (HIRMAb-IDUA) Fusion Protein, AGT-181 in Patients With Mucopolysaccharidosis I (MPS I, Hurler Syndrome)
Brief Title: Safety and Dose Ranging Study of Human Insulin Receptor MAb-IDUA Fusion Protein in Adults and Children With MPS I
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ArmaGen, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AGT-181-101
Record Dates: First submitted 2017-02-09; First posted 2017-02-14 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Mucopolysaccharidosis I
Keywords: MPS I; Hurler Syndrome
MeSH Terms: conditions — Mucopolysaccharidosis I | interventions — valanafusp alpha

STUDY DESIGN:
Intervention Model Description: Stage 1: 6 adults will be given a single dose, assigned to 0.3, 1.0 or 3.0 mg/kg (with cohort assignment based on order of study entry)
  Stage 2: up to 15 children will be given repeat weekly doses for 26 weeks, assigned to 1.0, 3.0 and 6.0 or 9.0 mg/kg (with cohort assignment based on order of study entry). Early term
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stage 1 (adult) (Experimental): AGT-181
  Interventions: Drug: AGT-181
- Stage 2 (children) (Experimental): AGT-181
  Interventions: Drug: AGT-181

INTERVENTIONS:
Drug: AGT-181 — Human Insulin Receptor Monoclonal Antibody-Human alpha-L-iduronidase (HIRMAb-IDUA) Fusion Protein

SUMMARY:
AGT-181 is a fusion protein containing alpha-L-iduronidase that is intended to deliver the enzyme peripherally and to the brain, when administered intravenously. This is a safety and tolerability study to obtain safety and exposure data as well as information on the biological activity of the investigational drug.

This is a two-stage, sequential, single and multi-dose study of AGT-181 in patients with MPS I. The first stage will be an open-label, single-dose, dose-escalation cohort study and the second stage will be an open-label, multi dose, adaptive dose escalation cohort study.

DETAILED DESCRIPTION:
Stage 1:

Stage one will be a single-dose, dose-escalation study in cohorts of 2 patients with Hurler-Scheie or Scheie syndrome age 18 or greater who have not had ERT for at least 7 days prior to starting treatment. Approximately 3 cohorts will be enrolled sequentially, with safety data from the previous cohort being reviewed prior to escalation to the next higher dose cohort. Patients will be assigned to cohorts on the basis of their order of entry into the study.

The first cohort will be administered a single intravenous infusion of 0.3 mg/kg AGT-181 diluted in D5 normal saline over 4 hours. All patients will be observed for safety for 28 days after dosing. For dose escalation, the decision to proceed to a higher dose of AGT-181 will be made by the Sponsor and the investigator(s) after review of the available safety and tolerability data on or after 7 days post dose from patients who received the previous dose.

Dose escalation to a higher dose cohort can occur providing there are no dose limiting toxicities (DLT), defined as Grade 3 (severe or medically significant but not immediately life threatening) or higher adverse event according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03

Stage 2:

Assuming safety and tolerability in Stage 1, a second stage will be initiated using a multi-dose, safety, tolerability and proof of concept effect design in children (age 2 or older) with Hurler or Hurler-Scheie with CNS involvement who are either ERT naïve or will have not received ERT for at least 7 days prior to first dose of AGT-181.

This second stage of the study will be conducted in dose groups of up to 5 patients per group who will receive AGT-181; it is planned that up to 10 patients will be enrolled (2 dose cohorts). Additional patients or cohorts may be enrolled in order to evaluate specific safety or PK issues or if it is felt that an active dose has not yet been reached. If an active dose is not achieved, an additional cohort of 5 patients will be enrolled at a higher dose of AGT-181, A maximum of 15 patients will be enrolled in stage 2. These cohorts will be studied in staggered fashion with safety and efficacy data from the previous cohort being reviewed as part of the decision to commence treatment in additional cohorts. Patients will be assigned to cohorts on the basis of their order of entry into the study.

The first cohort will be administered a dose one level below the maximum tolerated (MTD) or maximum administered dose (MAD) from the single dose stage 1 (ie. if the MTD is 3.0 mg/kg from Stage 1 than the starting dose in this stage will be 1.0 mg/kg). AGT-181 will be administered as a once weekly intravenous infusion in D5 normal saline over 4 hours for the first eight infusions. Depending upon tolerability, the rate may be increased to be administered over 1-4 hours. Investigators are permitted to use their clinical judgment and standard protocols in determining whether to administer pre-infusion medications such as antihistamines and antipyretics. In cases where the patient has had a previous infusion reaction(s) to ERT, then premedication should be given prior to each infusion per clinical site standard protocol.

For dose escalation, the decision to proceed to a higher dose of AGT-181 will be made by the Sponsor and the investigator(s) after review of the available safety and tolerability data from patients who received the previous dose.

Dose escalation to a higher dose cohort can occur providing there is no dose limiting toxicity (DLT) in the first 3 patients treated for 28 days or more. If one patient of 3 develops a DLT, then dose escalation may not occur until the remaining 2 patients have completed 28 days of dosing and there have been no further DLTs. A DLT is defined as a Grade 3 (severe or medically significant but not immediately life threatening) or higher adverse event according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.

If a Grade 3 or worse event is clearly attributable to a non-treatment event and therefore not a suspected adverse reaction: [21CFR312.32(a)] (for example, trauma secondary to an accident, or spurious lab value not confirmed on repeat) the event will not be considered a DLT for dose escalation purposes after review and agreement by both the Sponsor's Medical Monitor and Principal Investigator.

In addition to adverse events occurring during the first 28 days, late and chronic toxicities will be evaluated and taken into account in determining the safety of each dose level for future studies and the need for additional cohorts in this study.

ELIGIBILITY:
Inclusion Criteria:

* Written consent and assent as required
* Diagnosis of MPS 1 confirmed by clinical signs and symptoms, documented fibroblast or leukocyte IDUA enzyme activity of less than 10% the lower limit of normal
* Female patients must not be pregnant, willing to utilize appropriate birth control methods and undergo pregnancy testing during the study
* if taking standard ERT, must be willing to discontinue for 1 week prior to dosing and for the study duration

Additional Inclusion Criteria, Stage 1:

* 18 years of age or older
* must have a diagnosis of Hurler-Scheie or Scheie syndrome

Additional Inclusion Criteria, Stage 2:

* 2 years of age or older (and less than 18)
* must be willing to undergo CNS testing, including assessment of CSF via lumbar puncture, MRI scans and neurocognitive testing
* must have evidence of Hurler-Scheie or Scheie with CNS involvement, as evidence by:
* score of 1 to 3 standard deviations below mean on IQ testing (i.e. IQ=55 or more) or in one domain of neuropsychological function (language, memory, non-verbal ability) OR
* documented historical evidence of a decline greater than 1 standard deviation on sequential testing, OR
* score between 0.75 and 1 standard deviation below the mean, AND cognitive deficit affects daily performance

Exclusion Criteria:

* Refusal to complete all assessments
* Pregnant or Lactating
* Received investigational drug within 1 year prior to study enrollment
* Medical condition or extenuating circumstance that, in the opinion of the investigator, may interfere with study compliance
* CSF pressure greater than 25 cm H20 (18 mm Hg)
* Known hypersensitivity to alpha-L-iduronidase (IDUA/Aldurazyme) or any components/excipients found in AGT-181
* Previous successful (engrafted) hematopoietic stem cell transplantation which has resulted in normalization of urinary glycosaminoglycans (GAGs); or major organ transplantation
* Clinically significant spinal cord compression or evidence of cervical instability (i.e. expected to require intervention during study participation)
* History of diabetes mellitus or hypoglycemia

Additional Exclusion Criteria, Stage 2:

* Has ventriculoperitoneal shunt
* IQ below 55
* Previously received AGT-181 in Stage 1 of the study

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Stage 1: number of patients with adverse events as a measure of safety and tolerability of a single dose | 4 weeks
Stage 2: number of patients with adverse events as a measure of safety and tolerability of repeat weekly doses | 26 weeks

SECONDARY OUTCOMES:
PK parameters (maximal concentration, half-life, AUC, distribution and clearance) of AGT-181 | 26 weeks
change in total urinary glycosaminoglycans (GAGs) | 26 weeks
change in functional capacity (6-minute walk test) or lung function (forced vital capacity) | 26 weeks
change in shoulder range of motion (ROM) | 26 weeks
change in liver and/or spleen volume (measured by MRI) | 26 weeks

OTHER OUTCOMES:
change in levels of heparan sulfate and/or dermatan sulfate in cerebrospinal fluid (CSF) | 26 weeks
change in levels of heparan sulfate and/or dermatan sulfate in plasma | 26 weeks
change in neurocognition (measured by VABS-II and BSID-III or KABC-II) | 26 weeks
change in CNS neuroimaging (brain volumetric MRI and diffusion tensor imaging, DTI) | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Patrice P Rioux, MD PhD, Study Director — ArmaGen, Inc
Locations (1):
- HCPA - Hospital das Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Giugliani R, Giugliani L, de Oliveira Poswar F, Donis KC, Corte AD, Schmidt M, Boado RJ, Nestrasil I, Nguyen C, Chen S, Pardridge WM. Neurocognitive and somatic stabilization in pediatric patients with severe Mucopolysaccharidosis Type I after 52 weeks of intravenous brain-penetrating insulin receptor antibody-iduronidase fusion protein (valanafusp alpha): an open label phase 1-2 trial. Orphanet J Rare Dis. 2018 Jul 5;13(1):110. doi: 10.1186/s13023-018-0849-8. PMID 29976218